CLINICAL TRIAL: NCT05947227
Title: Effects of BBT Versus Diaphragmatic Breathing on Exercise Capacity and Quality of Life in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0311
Record Dates: First submitted 2023-06-14; First posted 2023-07-17 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Breathing Technique
Keywords: Chronic obstructive pulmonary disease/COPD; Diaphragmatic breathing technique
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Group A will be treated with manual chest physical therapy and Buteyko breathing technique Group-B will be treated with manual chest physical therapy and Diaphragmatic breathing technique. Patients will perform the technique 5 times a weeks for 8weeks and treatment evaluation will be done after 8 weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual chest physical therapy and Buteyko breathing technique (Experimental): Group A will be treated with manual chest physical therapy and Buteyko breathing technique
  Interventions: Other: Buteyko breathing technique
- manual chest physical therapy and Diaphragmatic breathing technique. (Experimental): Group-B will be treated with manual chest physical therapy and Diaphragmatic breathing technique.
  Interventions: Other: Diaphragmatic breathing technique.

INTERVENTIONS:
Other: Buteyko breathing technique — Group A : will be treated with manual chest physiotherapy & Buteyko Breathing exercise
  Arms: manual chest physical therapy and Buteyko breathing technique
Other: Diaphragmatic breathing technique. — Group B : will be treated with manual chest physiotherapy & Diaphragmatic Breathing Treatment evaluation will be done after 8 weeks through 6MWT & St George respiratory Questionnaire. Patients will perform technique 5 times a weeks for 8 weeks
  Arms: manual chest physical therapy and Diaphragmatic breathing technique.

SUMMARY:
Group A will be treated with manual chest physical therapy and Buteyko breathing technique Group-B will be treated with manual chest physical therapy and Diaphragmatic breathing technique. Patients will perform the technique 5 times a weeks for 8weeks and treatment evaluation will be done after 8 weeks

DETAILED DESCRIPTION:
A randomized clinical trial will be conducted at Gulab Devi Hospital, Lahore through convenience sampling technique on 48 patients which will be allocated through simple random sampling through sealed enveloped into group A and group B. Pre-treatment values of patients exercise capacity will be recorded by 6MWT/6MWD- 6 minute walk test/ 6 minutes' walk distance and patients quality of life through St George respiratory questionnaire as primary outcomes while oxygen saturation, heart rate will be measured by pulse oximtery during 6MWT as secondary outcomes. Group A will be treated with manual chest physical therapy and Buteyko breathing technique Group-B will be treated with manual chest physical therapy and Diaphragmatic breathing technique. Patients will perform the technique 5 times a weeks for 8weeks and treatment evaluation will be done after 8 weeks.

Data will be analyzed using SPSS software version 25.After assessing normality of data by Shapiro-Wilk test , it will be decidedeither parametric or non-parametric test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age group : 40-65 years
* Both males and females
* Clinical diagnosis of COPD confirmed by smoking history and PFT airflow
* Patients taking their regular medications e.g bronchodilator

Exclusion Criteria:

* Restrictive lung disease
* Pneumothorax
* Resting O2 saturation <90% with room air breathing
* Recent exacerbations
* Patients with active viral or bacterial infection
* Abdominal or thoracic surgery (<3months ago)
* Cardiologic conditions (<6months ago e.g Myocardial infarction or unstable angina
* Intubated Patients
* Orthopedic or urogenital conditions
* Neurological disorders limiting cognition & mobility

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Distance | 4 weeks.
  Distance will be measured in meter through 6 minute walk test.

SECONDARY OUTCOMES:
St George Respiratory Questionnaire for quality of life : | 4 weeks.
  St George Respiratory Questionnaire/SGRQ is a well established disease specific for health status in asthma and COPD (26).A total three component scores are provided , symptoms (8 items) , activity (16 items) and impacts (26 items), 50 items vary as likert type scale and dichotomus (true/false). In the symptom component , patients are instructed to recall their symptoms in a specific time frame of 1 month , 3 months or 1 year. Other items are not time specific.Scores ranged from 0 ( no impairment ) to 100 ( worst health status)

OTHER OUTCOMES:
oxygen saturation | 4 weeks
  Oxygen saturation will be measured through pulse oximeter.
heart rate | 4 weeks
  Pulse rate will be measured through pulse oximeter which will be consider as heart rate of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Faisal, MS.CPPT, Principal Investigator — Riphah International University
Locations (1):
- Gulab Devi Hospital, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iheanacho I, Zhang S, King D, Rizzo M, Ismaila AS. Economic Burden of Chronic Obstructive Pulmonary Disease (COPD): A Systematic Literature Review. Int J Chron Obstruct Pulmon Dis. 2020 Feb 26;15:439-460. doi: 10.2147/COPD.S234942. eCollection 2020. PMID 32161455
- [Background] Chatreewatanakul B, Othaganont P, Hickman RL. Early symptom recognition and symptom management among exacerbation COPD patients: A qualitative study. Appl Nurs Res. 2022 Feb;63:151522. doi: 10.1016/j.apnr.2021.151522. Epub 2021 Nov 6. PMID 35034709
- [Background] Adeloye D, Song P, Zhu Y, Campbell H, Sheikh A, Rudan I; NIHR RESPIRE Global Respiratory Health Unit. Global, regional, and national prevalence of, and risk factors for, chronic obstructive pulmonary disease (COPD) in 2019: a systematic review and modelling analysis. Lancet Respir Med. 2022 May;10(5):447-458. doi: 10.1016/S2213-2600(21)00511-7. Epub 2022 Mar 10. PMID 35279265
- [Background] Gea J, Agusti A, Roca J. Pathophysiology of muscle dysfunction in COPD. J Appl Physiol (1985). 2013 May;114(9):1222-34. doi: 10.1152/japplphysiol.00981.2012. Epub 2013 Mar 21. PMID 23519228
- [Background] Cavalcanti JD, Fregonezi GAF, Sarmento AJ, Bezerra T, Gualdi LP, Pennati F, Aliverti A, Resqueti VR. Electrical activity and fatigue of respiratory and locomotor muscles in obstructive respiratory diseases during field walking test. PLoS One. 2022 Apr 1;17(4):e0266365. doi: 10.1371/journal.pone.0266365. eCollection 2022. PMID 35363800
- [Background] Tang CY, Taylor NF, Blackstock FC. Chest physiotherapy for patients admitted to hospital with an acute exacerbation of chronic obstructive pulmonary disease (COPD): a systematic review. Physiotherapy. 2010 Mar;96(1):1-13. doi: 10.1016/j.physio.2009.06.008. Epub 2009 Sep 22. PMID 20113757
- [Background] Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Chen R, Decramer M, Fabbri LM, Frith P, Halpin DM, Lopez Varela MV, Nishimura M, Roche N, Rodriguez-Roisin R, Sin DD, Singh D, Stockley R, Vestbo J, Wedzicha JA, Agusti A. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report. GOLD Executive Summary. Am J Respir Crit Care Med. 2017 Mar 1;195(5):557-582. doi: 10.1164/rccm.201701-0218PP. PMID 28128970